CLINICAL TRIAL: NCT03463044
Title: A Phase I, Randomised, Placebo Controlled Study to Assess the Safety, Tolerability and Pharmacokinetic Profiles of Ascending, Single, Intravenous Doses of MOTREM (LR12) in Healthy Male Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic Profiles of MOTREM (LR12) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inotrem (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MOT-C-104
Record Dates: First submitted 2018-02-27; First posted 2018-03-13 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — nangibotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo
- MOTREM 1 (Experimental): nangibotide dose 1
  Interventions: Drug: nangibotide
- MOTREM 2 (Experimental): Nangibotide dose 2
  Interventions: Drug: nangibotide
- MOTREM 3 (Experimental): Nangibotide dose 3
  Interventions: Drug: nangibotide
- MOTREM 4 (Experimental): Nangibotide dose 4
  Interventions: Drug: nangibotide
- MOTREM 5 (Experimental): Nangibotide dose 5
  Interventions: Drug: nangibotide
- MOTREM 6 (Experimental): Nangibotide dose 6
  Interventions: Drug: nangibotide
- MOTREM 7 (Experimental): Nangibotide dose 7
  Interventions: Drug: nangibotide
- MOTREM 8 (Experimental): Nangibotide dose 8
  Interventions: Drug: nangibotide

INTERVENTIONS:
Drug: nangibotide — Continous i.v. infusion
  Other Names: LR12; MOTREM
  Arms: MOTREM 1; MOTREM 2; MOTREM 3; MOTREM 4; MOTREM 5; MOTREM 6; MOTREM 7; MOTREM 8
Drug: Placebo — Placebo
  Other Names: matched placebo
  Arms: Placebo

SUMMARY:
This was a single center, randomized, placebo-controlled study with a sequential i.v. dose escalation cohorts design, to assess safety, tolerability and pharmacokinetics of MOTREM (nangibotide) in healthy volunteers

DETAILED DESCRIPTION:
This was a dose escalation study in healthy volunteers to evaluate the safety and pharmacokinetics of nangibotide in humans

ELIGIBILITY:
Inclusion Criteria:

* healthy male
* ≥18 to ≤45 years old
* Body mass index (BMI) between 18-30 kg/m² inclusive
* Written informed consent to participate.

Main Exclusion Criteria:

* Any clinically relevant acute or chronic diseases
* Any history of drug or alcohol abuse
* Any History of clinical significant disease as determined by medical history, physical examination or other evaluations.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2016-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Cuvier, Study Director — Inotrem
Locations (1):
- Richmond Pharmacology Ltd., Croydon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cuvier V, Lorch U, Witte S, Olivier A, Gibot S, Delor I, Garaud JJ, Derive M, Salcedo-Magguilli M. A first-in-man safety and pharmacokinetics study of nangibotide, a new modulator of innate immune response through TREM-1 receptor inhibition. Br J Clin Pharmacol. 2018 Oct;84(10):2270-2279. doi: 10.1111/bcp.13668. Epub 2018 Jul 20. PMID 29885068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the UK. The first subject first visit was on 01 April 2016 and last subject last visit was on 25 August 2016.
Pre-assignment Details: Subjects were screened within 14 days and screening could be performed over multiple days prior to entering the study on Day -1. A total of 27 subjects were randomized and 26 subjects completed the study (1 subject was lost to follow-up and was prematurely withdrawn).
Groups:
- 1 mg (Loading Dose) Nangibotide: Part A, Cohort 1: 1 mg (loading dose) over 15 minutes i.v.
- 10 mg (Loading Dose) Nangibotide: Part A, Cohort 2: 10 mg (loading dose) over 15 minutes i.v.
- 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide: Part B, Cohort 3: 0.5 mg/kg i.v. loading dose and 0.03 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
- 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide: Part B, Cohort 4: 1 mg/kg i.v. loading dose and 0.1 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
- 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide: Part B, Cohort 5: 2 mg/kg i.v. loading dose and 0.3 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
- 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide: Part B, Cohort 6: 5 mg/kg i.v. loading dose and 1 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
- 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide: Part B, Cohort 7: 5 mg/kg i.v. loading dose and 3 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
- 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide: Part B, Cohort 8: 5 mg/kg i.v. loading dose and 6 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
Period: Overall Study
Arm/Group | Placebo | 1 mg (Loading Dose) Nangibotide | 10 mg (Loading Dose) Nangibotide | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide
Started | 6 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 6 | 1 | 2 | 3 | 3 | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported in clinical study report according to the patients enrolled in each cohort, not separately for placebo and investigational medicinal product.
Groups:
- Cohort 1: 1 mg nangibotide over 15 minutes i.v.
- Cohort 2: 10 mg nangibotide over 15 minutes i.v.
- Cohort 3: 0.5 mg/kg i.v. and 0.03 mg/kg/h nangibotide i.v. over 7 hours and 45 min or placebo
- Cohort 4: 1 mg/kg i.v. and 0.1 mg/kg/h i.v. nangibotide over 7 hours and 45 min or placebo
- Cohort 5: 2 mg/kg i.v. and 0.3 mg/kg/h i.v. nangibotide over 7 hours and 45 min or placebo
- Cohort 6: 5 mg/kg i.v. and 1 mg/kg/h i.v. nangibotide over 7 hours and 45 min or placebo
- Cohort 7: 5 mg/kg i.v. and 3 mg/kg/h i.v. nangibotide over 7 hours and 45 min or placebo
- Cohort 8: 5 mg/kg i.v. and 6 mg/kg/h i.v. nangibotide over 7 hours and 45 min or placebo
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Total
Number analyzed (Participants) | 1 | 2 | 4 | 4 | 4 | 4 | 4 | 4 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 4 | 4 | 4 | 4 | 4 | 4 | 27
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 2 | 4 | 4 | 4 | 4 | 4 | 4 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3
  White | 1 | 2 | 4 | 1 | 3 | 4 | 3 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1 | 2 | 4 | 4 | 4 | 4 | 4 | 4 | 27
Weight [Median (Full Range); unit: kg] | 81.2 [81.2 to 81.2] | 68.6 [57.2 to 80] | 71.7 [65.3 to 75.5] | 77.1 [72.4 to 80.4] | 73.1 [61.4 to 100] | 74.4 [58.7 to 78.2] | 77.1 [70.6 to 84.9] | 76.7 [73.5 to 77.1] | 75.7 [57.2 to 100]
Height [Median (Full Range); unit: cm] | 189.0 [189.0 to 189.0] | 169.5 [166 to 173] | 178.0 [176 to 185] | 180.0 [164 to 186] | 183.0 [176 to 188] | 178.0 [173 to 182] | 179.5 [172 to 187] | 182.0 [175 to 189] | 180.0 [164 to 189]
BMI [Median (Full Range); unit: kg/m²] | 22.7 [22.7 to 22.7] | 23.7 [20.76 to 26.73] | 22.3 [20.15 to 23.82] | 24.2 [20.93 to 28.85] | 21.9 [18.74 to 29.22] | 23.5 [18.95 to 24.42] | 24.1 [21.08 to 27.41] | 23.1 [21.58 to 24.08] | 23.4 [18.74 to 29.22]

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability: the Number of Subjects Experiencing Treatment Emergent Adverse Events
Description: The number of subjects experiencing treatment emergent adverse events was collected to assess the safety and tolerability of MOTREM (LR12) in comparison with placebo.
Time Frame: 30-44 days
Measure: Count of Participants; unit: Participants
Groups:
- 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose): Part B, Cohort 8: 5 mg/kg i.v. loading dose and 6 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
Arm/Group | Placebo | 1 mg (Loading Dose) Nangibotide | 10 mg (Loading Dose) Nangibotide | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose)
Number analyzed (Participants) | 6 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1

2. Secondary Outcome: Pharmacokinetics (Maximum Plasma Concentration)
Description: Plasma concentrations of LR12 were measured by a validated liquid chromatography-mass spectrometry (LC-MS/MS) assay and analyzed using noncompartmental methods to obtain estimates of the pharmacokinetic parameter of Maximum Plasma Concentration (Cmax).
Time Frame: Maximum Plasma Concentration (Cmax) was assessed only for Groups 3-8 who received loading dose over 15 min and maintenance dose over 7 h and 45 min. Cmax is determined over a period of time starting from predose to 10h after start of the loading dose.
Population: In cohort 1 and cohort 2, there was 1 subject per cohort and the subjects received only a loading dose. LR12 plasma concentrations were quantifiable only at 15 min post-start of the infusion. For this reason, no PK analysis was performed for these two cohorts and for this reason results were not presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
ng/mL | 256.20 (39) | 638.04 (25) | 1643.25 (22) | 3818.94 (1) | 4185.47 (66) | 4200.05 (21)

3. Secondary Outcome: Statistical Analysis of LR12 PK Parameters: Steady State Concentration During the Maintenance Infusion (Cavg30-465)
Description: Plasma concentrations of LR12 were measured by a validated LC-MS/MS assay and analyzed using noncompartmental methods to obtain estimates of the PK parameter of steady state concentration during the maintenance infusion (Cavg30-465).
Time Frame: Cavg30-465 was assessed only for Groups 3-8 who received loading dose over 15 min and maintenance dose over 7 h and 45 min. Cavg30-465 is determined over a period of time starting from predose to 10h after start of the loading dose.
Population: In cohort 1 and cohort 2, there was 1 subject per cohort and the subjects received only a loading dose. LR12 plasma concentrations were quantifiable only at 15 min post-start of the infusion. For this reason, no PK analysis was performed for these two cohorts. For Cohort 3 values for Cavg30-465 were non-calculable. Hence, the results for Cohorts 1,2 and 3 are not presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose): Part B, Cohort 6: 5 mg/kg i.v. loading dose and 1 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
- 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose): Part B, Cohort 7: 5 mg/kg i.v. loading dose and 3 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
Arm/Group | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
ng/mL | NA (NA) — For Cohort 3 values for Cavg30-465 were non-calculable because of missing values for some of the 3 patients because below the level of detection | 13.46 (18) | 36.61 (14) | 152.41 (12) | 418.05 (22) | 983.19 (20)

4. Secondary Outcome: Statistical Analysis of LR12 PK Parameters: t1/2
Description: Plasma concentrations of LR12 were measured by a validated LC-MS/MS assay and analyzed using noncompartmental methods to obtain estimates of the PK parameter of terminal half-life (t1/2).
  Of note, apparent increase in half-life at increasing doses is explained by the detection of a slow elimination phase, which was below limit of quantification for the lower doses.
Time Frame: t1/2 was assessed only for Groups 3-8 who received loading dose over 15 min and maintenance dose over 7 h and 45 min. t1/2 is determined over a period of time starting from 7 h and 45 min to 10h after start of the loading dose (decaying period).
Population: Up to cohort 5, due to paucity of the data, t1/2 could not be determined, hence the results for these cohorts are not presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: minute
Groups:
- 0.5 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide: Part B, Cohort 4: 0.5 mg/kg i.v. loading dose and 0.1 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
- 0.5 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide: Part B, Cohort 5: 0.5 mg/kg i.v. loading dose and 0.3 mg/kg/h maintenance dose i.v. over 7 hours and 45 min
Arm/Group | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 0.5 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 0.5 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
minute | NA (NA) — Up to cohort 5, due to paucity of the data (below the level of detection), t1/2 could not be determined | NA (NA) — Up to cohort 5, due to paucity of the data (below the level of detection), t1/2 could not be determined. | NA (NA) — Up to cohort 5, due to paucity of the data (below the level of detection), t1/2 could not be determined. | 1.63 (20) | 17.87 (23) | 40.70 (76)

5. Secondary Outcome: Statistical Analysis of LR12 PK Parameters: AUC0-t
Description: Plasma concentrations of LR12 were measured by a validated LC-MS/MS assay and analyzed using noncompartmental methods to obtain estimates of the PK parameter of the area under the plasma concentration curve (h.ng/mL) from time zero (predose) to the time of last observed concentration (t) measured (which can go up to 10h post loading dose start) using a linear trapezoidal method (AUC0-t).
Time Frame: AUC0-t was assessed only for Groups 3-8 who received loading dose over 15 min and maintenance dose over 7 h and 45 min. AUC0-t is determined over a period of time starting time zero (predose) to the time of last observed concentration (t).
Population: There was 1 subject per cohort in cohort 1 and cohort 2 and the subjects received only a loading dose. LR12 (nangibotide) plasma concentrations were quantifiable only at 15 min post-start of the infusion. For this reason, no PK analysis was planned for these two cohorts and no results were presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/ml
Arm/Group | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
h.ng/ml | 101.98 (11) | 244.38 (14) | 661.60 (23) | 2153.14 (11) | 4208.65 (29) | 8556.69 (17)

6. Secondary Outcome: Statistical Analysis of LR12 PK Parameters: AUC0-∞
Description: Plasma concentrations of LR12 were measured by a validated LC-MS/MS assay and analyzed using noncompartmental methods to obtain estimates of the PK parameter of AUC0-∞.
  AUC0-∞ represents the area under the plasma concentration-time curve (h.ng/mL) from time 0 to infinity (AUC0- ∞= AUC0-t + [Ct/ke], where Ct = the observed concentration of drug for the last sample on the PK profile in which drug was detected, and ke represents the terminal rate constant). The percentage of extrapolation of AUC0-∞ should not exceed 20%.
Time Frame: AUC0-∞ was assessed only for Groups 3-8 who received loading dose over 15 min and maintenance dose over 7 h and 45 min. AUC0-∞ is determined over a period of time starting time zero (predose) to infinity (cf. extrapolation formula in the above section).
Population: The percentage of extrapolation of AUC0-∞ was below 1% in subjects up to cohort 5, and due to this it was not determined for these subjects. For this reason, results were not presented for cohorts 1-5.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/ml
Arm/Group | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 0.5 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 0.5 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
h.ng/ml | NA (NA) — The percentage of extrapolation of AUC0-∞ was below the level of detection of 1% in subjects up to cohort 5, and due to this it was not determined for these subjects. | NA (NA) — The percentage of extrapolation of AUC0-∞ was below the level of detection of 1% in subjects up to cohort 5, and due to this it was not determined for these subjects. | NA (NA) — The percentage of extrapolation of AUC0-∞ was below the level of detection of 1% in subjects up to cohort 5, and due to this it was not determined for these subjects. | 2153.38 (11) | 4211.90 (29) | 8565.30 (17)

7. Secondary Outcome: Statistical Analysis of LR12 PK Parameters: CL
Description: Plasma concentrations of LR12 were measured by a validated LC-MS/MS assay and analyzed using noncompartmental methods to obtain estimates of the PK parameter of systemic clearance (CL). The systemic clearance was estimated using the formula: CL = K0/ Css where K0 is the perfusion rate (ng/kg/h) and Css is the concentration at the end of perfusion (C at 465 min).
  Of note, this narrow range of the clearance values indicates that the apparent increases in t1/2 and volume of distribution as a function of doses are not due to a non-linearity in the pharmacokinetics, but to the limit of quantification of the bioanalytical assay.
Time Frame: CL was assessed only for Groups 3-8 who received loading dose over 15 min and maintenance dose over 7 h and 45 min (465 min). CL is calculated based on the perfusion rate (ng/kg/h) and the concentration at the end of perfusion (7h45min = 465min).
Population: There was 1 subject per cohort and the subjects received only a loading dose in cohort 1 and cohort 2. LR12 (nangibotide) plasma concentrations were quantifiable only at 15 min post-start of the infusion. No PK analysis was planned for these two cohorts. Also, CL values for cohort 3 were non-calculable. For this reason, results for cohorts 1-3 are not presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg/h
Arm/Group | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
L/kg/h | NA (NA) — CL values for cohort 3 were non-calculable due to very low LR12 concentration at 7h45min post maintenance dose (below the level of detection) | 9.47 (9) | 6.79 (17) | 6.73 (25) | 5.66 (22) | 7.50 (20)

8. Secondary Outcome: Statistical Analysis of LR12 PK Parameters: Volume of Distribution (V)
Description: The volume of distribution was estimated according to the following equation: V= CL x MRT (mean residence time). However, regarding administration procedures, MRT could not be calculated precisely. Furthermore, in some cases MRT could not be estimated. Thus, the following formula was used V = CL / ke.
  The terminal rate constant (ke) was estimated by log-linear regression analysis on data points visually assessed to be on the terminal log-linear phase.
  Of note, it can be said that this apparent increase in V is also explained by the detection of a slow elimination phase, which was below limit of quantification for the lower doses.
Time Frame: V was assessed only for Groups 3-8 who received loading dose over 15 min and maintenance dose over 7 h and 45 min. V is derived from both CL and ke which are calculated from the LR12 concentration time curve from predose to 10h after loading dose start.
Population: There was 1 subject per cohort In cohort 1 and cohort 2 and the subjects received only a loading dose. LR12 plasma concentrations were quantifiable only at 15 min post-start of the infusion. No PK analysis was planned for these two cohorts. Also, V values for cohort 3, 4 and 5 were non-calculable. For this reason, no results were presented for cohorts 1-6.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 0.5 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 0.5 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
L/kg | NA (NA) — V values for cohort 3, 4 and 5 were non-calculable (below the level of detection). | NA (NA) — V values for cohort 3, 4 and 5 were non-calculable (below the level of detection). | NA (NA) — V values for cohort 3, 4 and 5 were non-calculable (below the level of detection). | 0.26 (46) | 2.43 (30) | 7.34 (62)

9. Secondary Outcome: Statistical Analysis of LR12 PK Parameters: Tmax
Description: Plasma concentrations of LR12 were measured by a validated LC-MS/MS assay and analysed using noncompartmental methods to obtain estimates of the PK parameter of the time at which Cmax is apparent, identified by inspection of the plasma drug concentration vs.time data by WinNonlin (tmax).
Time Frame: tmax was assessed only for Groups 3-8 who received loading dose over 15 min and maintenance dose over 7 h and 45 min. tmax is determined over a period of time starting from predose to 10h after start of the loading dose.
Population: There was 1 subject per cohort in cohort 1 and 2 and the subjects received only a loading dose. LR12 plasma concentrations were quantifiable only at 15 min post-start of the infusion. No PK analysis was planned for these two cohorts. For this reason, results for cohort 1 and 2 were not presented.
Measure: Median (Full Range); unit: minute
Arm/Group | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
minute | 15 [15 to 15] | 15 [15 to 15] | 15 [15 to 15] | 15 [15 to 15] | 5 [5 to 15] | 5 [5 to 15]

10. Secondary Outcome: Statistical Analysis of LR12 PK Parameters: t Last
Description: This PK parameter was calculated from measured plasma concentrations of LR12 and it represents the time of last observed concentration.
Time Frame: t last was assessed only for Groups 3-8 who received loading dose over 15 min and maintenance dose over 7 h and 45 min. t last is determined as the time of last observed concentration which can go up to 10h after loading dose start.
Population: as for outcome 9
Measure: Median (Full Range); unit: minute
Arm/Group | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
minute | 465 [360 to 484] | 484 [484 to 493] | 484 [484 to 484] | 487 [487 to 487] | 510 [510 to 511] | 600 [510 to 601]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored until day 28 (end of study visit).
Description: All TEAEs were mild in severity, and considered unrelated to the study drug. There was no SAE and no TEAE leading to treatment stop.
Arm/Group | Placebo | 1 mg (Loading Dose) Nangibotide | 10 mg (Loading Dose) Nangibotide | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide | 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide | 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/1 | 0/2 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/1 | 0/2 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/6 | 0/1 | 1/2 | 1/3 | 1/3 | 0/3 | 0/3 | 1/3 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | 1 mg (Loading Dose) Nangibotide (N=1) | 10 mg (Loading Dose) Nangibotide (N=2) | 0.5 mg/kg (Loading Dose) and 0.03 mg/kg/h (Maintenance Dose) Nangibotide (N=3) | 1 mg/kg (Loading Dose) and 0.1 mg/kg/h (Maintenance Dose) Nangibotide (N=3) | 2 mg/kg (Loading Dose) and 0.3 mg/kg/h (Maintenance Dose) Nangibotide (N=3) | 5 mg/kg (Loading Dose) and 1 mg/kg/h (Maintenance Dose) Nangibotide (N=3) | 5 mg/kg (Loading Dose) and 3 mg/kg/h (Maintenance Dose) Nangibotide (N=3) | 5 mg/kg (Loading Dose) and 6 mg/kg/h (Maintenance Dose) Nangibotide (N=3)
Cerumen removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03463044/Prot_SAP_000.pdf